CLINICAL TRIAL: NCT04557020
Title: Adding Neoadjuvant and Adjuvant PD-1 Inhibitor to Neoadjuvant Chemotherapy Plus Concurrent Chemoradiotherapy in the Treatment of High-risk Nasopharyngeal Carcinoma
Brief Title: Adding PD-1 Inhibitor to Neoadjuvant and Adjuvant for NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC2020-001
Record Dates: First submitted 2020-09-02; First posted 2020-09-21 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — spartalizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): IC with anti-PD1 mab+CCRT+anti-PD1 mab
  Interventions: Drug: PD-1 antibody; Drug: Gemcitabine; Drug: Cisplatin; Radiation: IMRT
- Arm B (Active Comparator): IC+CCRT
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: PD-1 antibody — neoadjuvant: PD-1 inhibitor Toripalimab 240mg combined with neoadjuvant chemotherapy by cis Platinum and gemcitabine every 3 weeks for 3 cycles ; adjuvant: Toripalimab 240mg every 3 weeks for 9 cycles after concurrent chemoradiotherapy
  Arms: Arm A
Drug: Gemcitabine — neoadjuvant chemotherapy: 1000mg/m2 in day 1 and day 8 and repeats every 3 weeks for 3 cycles
Drug: Cisplatin — neoadjuvant chemotherapy: 80mg/m2 in day 1, and repeats every 3 weeks for 3 cycles. Concurrent chemoradiotherapy: Cisplatin 100mg/m2 in day 1, 22, and 43 during IMRT
Radiation: IMRT — 70Gy to GTV, 60Gy to CTV1 and 54Gy to CTV2 in 32 to 33 fractions

SUMMARY:
This is a randomized clinical trial comparing neoadjuvant and adjuvant PD-1 inhibitor Toripalimab plus neoadjuvant chemotherapy and concurrent chemoradiotherapy versus neoadjuvant chemotherapy and concurrent chemoradiotherapy alone in high-risk nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma
2. Clinical staged as T4 or N3 （according to the 8th AJCC edition）
3. No evidence of distant metastasis (M0)
4. Male and no pregnant female
5. ECOG (Eastern Cooperative OncologyGroup) scale 0-1
6. WBC ≥ 4×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
7. Normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN)
8. Normal renal function test ( creatinine clearance ≥60 ml/min)

Exclusion Criteria:

1. Recurrent or distant metastatic disease.
2. History of malignant tumors (except cured basal cell carcinoma or uterine cervical carcinoma in situ) within the last 5 years.
3. History of radiotherapy or chemotherapy.
4. History of immunodeficiency disease
5. History of organ transplantation
6. Presence of life-threatening illness
7. Uncontrolled hypercalcemia
8. Severe uncontrolled medical conditions or active infectious diseases
9. Use of large doses of glucocorticoids, anti-cancer monoclonal antibodies, or other immunosuppressive agents within 4 weeks.
10. Pregnant or breastfeeding female
11. Emotional disturbance or mental illness
12. Refusal or inability to sign informed consent

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 year
  From date of randomization to date of first documentation of progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 year
  From date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Distant Metastasis-Free Survival (DMFS) | 3 year
  From date of randomization to date of first documentation of distant metastases or until the date of the last followup visit.
Locoregional Relapse-Free Survival (LRRFS) | 3 year
  From date of randomization to date of first documentation of locoregional relapse or until the date of the last follow-up visit.
Objective Response Rate （ORR） | within 3 weeks after neoadjuvant treatment and 3 months after concurrent chemoradiotherapy
  Either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
adverse events (AEs) | 3 year
  Treatment-related AEs (trAEs) and immune-related AEs (irAEs) according to the Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jingao Li, M.D., Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (7):
- China (7):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Suizhou Central Hospital, Suizhou, Hubei
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - First Affiliated hospital of Gannan Medical University, Guangzhou, Jiangxi
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Pingxiang Peoples' Hospital, Pingxiang, Jiangxi

IPD SHARING:
Plan to Share IPD: No